CLINICAL TRIAL: NCT07207122
Title: Effects of Transcranial Ultrasound Stimulation (TUS) on Neurological and Cognitive Outcomes in Neurodegenerative Diseases.
Acronym: NDD-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanmai Technologies PBC dba Sanmai (Industry)
Collaborators: Acacia Research (Unknown); University of New Mexico (Other); BrainMind (Unknown); The Regenesis Project (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeurodegenerativeDisorders-01
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Parkinson's Disease (PD); Parkinson's Disease Dementia (PDD); Parkinson's Disease Dementia; Alzheimer's; Alzheimer's Disease (AD); Mild Cognitive Impairment
Keywords: Alzheimer's; Parkinson's; Low-intensity focused ultrasound neuromodulation; noninvasive neuromodulation; mild cognitive impairment; Parkinson's disease dementia
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open label transcranial focused ultrasound neuromodulation (Experimental): We will target a brain region involved in disease pathology.
  Interventions: Device: Transcranial focused ultrasound modulation administered to a region involved in disease pathology.

INTERVENTIONS:
Device: Transcranial focused ultrasound modulation administered to a region involved in disease pathology. — Using Sanmai's device to administer tFUS to regions of interest.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of transcranial focused ultrasound neuromodulation in improving neural function, cognitive and behavioral performance, and quality of life for patients with neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years

Ability to read and understand English

Clinical diagnosis of Alzheimer's, Parkinson's, Parkinson's dementia, mild cognitive impairment

Normal or corrected to normal vision and hearing

Must be medically stable as determined by investigators

Exclusion Criteria:

History of significant neurological disorders unrelated to the target disease

Implanted medical devices or metal implants incompatible with TUS or MRI

Uncontrolled heart or cardiac conditions or implants: severe arrhythmia, myocardial infarction, arterial angina

Psychiatric Conditions: individuals diagnosed with obsessive-compulsive disorder, psychosis, and/or bipolar disorder. Final eligibility will be determined after a thorough evaluation by the study clinicians.

Brain surgery, history of significant brain injury, seizures, or drug use deemed likely to interfere with participant safety or the experiment

Medications or drugs: A comprehensive review of current medications will be conducted by the study team. Medications known to significantly increase the risk of seizures or interact with study interventions will be carefully evaluated for safety. Final decisions on eligibility regarding medication use will be made by the study clinicians and/or PIs.

No other recreational drug use for at least 1 month prior to first treatment session

History of epilepsy: the prospective participant has had multiple seizures. If they have had one febrile seizure, provoked seizure, or acute symptomatic seizure, they may be included.

Current pregnancy

History of migraines (more than 4 days per month in the last 3 months)

Initiation of new neuromodulation or pharmacological treatment with last 6 weeks

Current cancer, or less than 5 years of remission from cancer

Weight over 350 lbs

Uncorrected hearing or visual impairment

Ingests more than 150mg of nicotine a day

Drug or alcohol addiction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Finger Tapping | 2 weeks
  A simple motor assessment used to measure speed, rhythm, and coordination of repetitive finger movements.
10-meter Timed Walk | 2 weeks
  A simple gait assessment in which a person is asked to walk 10 meters at a comfortable or maximum pace while the time taken is recorded. The test provides objective measures of walking speed and mobility.
Archimedes Spiral Test | 2 weeks
  A motor assessment in which a person is asked to draw a spiral on paper or a touchscreen. The accuracy, smoothness, and steadiness of the drawing provide a measure of tremor severity, fine motor control, and coordination.
PDQ-39 | 2 weeks
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a standardized self-report measure of health-related quality of life in people with Parkinson's disease. It includes 39 questions across eight domains-such as mobility, daily living, emotional well-being, stigma, and social support-providing a comprehensive view of how the condition impacts everyday life.
GAD-7 | 2 weeks
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is a brief self-report questionnaire used to screen for and assess the severity of anxiety symptoms. It is widely applied in both clinical practice and research to monitor treatment outcomes and track changes over time.
Beck Depression Inventory | 2 weeks
  The Beck Depression Inventory is a widely used self-report questionnaire that measures the presence and severity of depressive symptoms. It includes a series of multiple-choice items covering mood, cognitive patterns, and physical symptoms, making it useful for both clinical assessment and research.

SECONDARY OUTCOMES:
Finger Tapping | 1 month
  A simple motor assessment used to measure speed, rhythm, and coordination of repetitive finger movements.
10-meter timed walk test | 1 month
  A simple gait assessment in which a person is asked to walk 10 meters at a comfortable or maximum pace while the time taken is recorded. The test provides objective measures of walking speed and mobility.
Archimedes Spiral Test | 1 month
  A motor assessment in which a person is asked to draw a spiral on paper or a touchscreen. The accuracy, smoothness, and steadiness of the drawing provide a measure of tremor severity, fine motor control, and coordination.
PDQ-39 | 1 month
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a standardized self-report measure of health-related quality of life in people with Parkinson's disease. It includes 39 questions across eight domains-such as mobility, daily living, emotional well-being, stigma, and social support-providing a comprehensive view of how the condition impacts everyday life.
GAD-7 | 1 month
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is a brief self-report questionnaire used to screen for and assess the severity of anxiety symptoms. It is widely applied in both clinical practice and research to monitor treatment outcomes and track changes over time.
Beck Depression Inventory | 1 month
  The Beck Depression Inventory is a widely used self-report questionnaire that measures the presence and severity of depressive symptoms. It includes a series of multiple-choice items covering mood, cognitive patterns, and physical symptoms, making it useful for both clinical assessment and research.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Sanguinetti, PhD, Principal Investigator — Sanmai Technologies, PBC
Locations (1):
- The Regenesis Project, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared for analytics and improvements to the technologies.